CLINICAL TRIAL: NCT04800445
Title: Salivary C-reactive Protein,Mean Platelet Volume and Neutrophil Lymphocyte Ratio as Diagnostic Markers for Neonatal Sepsis
Brief Title: Salivary C- Reactive Protein, Mean Platelet Volume and Neutrophil Lymphocyte Ratio as Diagnostic Markers for Neonatal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eslam Mohamed Naeim, Emergency medicine and traumatology resident in sharq el madina hospital, Cairo University
Other Study IDs: MS-53-2020
Record Dates: First submitted 2021-02-26; First posted 2021-03-16 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group of fullterm neonates with neonatal sepsis
  Interventions: Diagnostic Test: Salivary CRP
- Healthy fullterm neonates
  Interventions: Diagnostic Test: Salivary CRP

INTERVENTIONS:
Diagnostic Test: Salivary CRP — Salivary C reactive protein in neonatal sepsis

SUMMARY:
To evaluate reliability of salivary C-reactive protein ,mean platelet volume , neutrophil -lymphocyte ratio , and platelet lymphocyte ratio in diagnosis of neonatal sepsis

ELIGIBILITY:
Inclusion Criteria:

* - Full term neonates of both genders from birth to the 28th day of life diagnosed with sepsis by history, clinical findings, laboratory findings, and blood culture. The clinical findings included the presence of three or more of the following:
* (1) temperature instability (hypothermia, hyperthermia) .
* (2) respiratory alterations (grunting, intercostal retractions, apnea, tachypnea, cyanosis) .
* (3) cardiovascular alterations (bradycardia, tachycardia, poor perfusion, hypotension) .
* (4) neurologic alterations (hypotonia, lethargy, seizures)
* (5) gastrointestinal alterations (feeding intolerance, abdominal distension). CRP values >10 mg/L were considered to be positive.

Exclusion Criteria:

* - Preterm neonates .
* Neonates with CNS malformations, metabolic disorders, chromosomal abnormalities, intrauterine growth restriction, or birth asphyxia were excluded from the study

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Full term neonates of both genders from birth to the 28th day of life who were admitted to Cairo University NICU with clinical features of either early- or late-onset neonatal sepsis diagnosed by culture, CRP more than 10 ,and has three or more the clinical findings of sepsis were enrolled in this study.
  Neonates with no symptoms or signs suggestive 0f sepsis who had been hospitalized In Cairo University Nicu . Serum CRP level for neonates in this group was negative (CRP < 10 mg/L) as control group.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2022-01-10 (Estimated)

PRIMARY OUTCOMES:
Salivary c reactive protein in neonatal sepsis | 28 days
  Salivary C reactive protein of value as non invasive procedure in diagnosis of neonatal sepsis

SECONDARY OUTCOMES:
Mean platelet volume | 28 days
  Asses the validity of Mean Platlet Volume as marker of neonatal sepsis which is equal about ( 9 - 11.4 ) in septic group and about ( 7.5 - 8.5 ) in control group

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo, Almanyal, Egypt